CLINICAL TRIAL: NCT07245277
Title: The Effect of Vitamin D Administration on Sepsis Score and C-Reactive Protein Levels in Preterm Infants With Neonatal Sepsis
Brief Title: Effect of Vitamin D as Adjuvant Therapy in Preterm Infants With Neonatal Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Michelle Angelica Wijaya, Principal Investigator, Fakultas Kedokteran Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DP. 04.03/D.XIV.6.5/337/2025
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Sepsis; Preterm Infants
Keywords: adjuvant therapy; neonatal sepsis; preterm infants; vitamin D
MeSH Terms: conditions — Neonatal Sepsis | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Antibiotics only (No Intervention): Group 1 consisted of subjects who were given only antibiotics due to medical conditions requiring fasting.
- Vitamin D 400 IU (Active Comparator): Group 2 consisted of subjects who were able to receive enteral nutrition, were given antibiotics, and were supplemented with vitamin D3 at a dose of 400 IU once daily for 7 days.
  Interventions: Drug: Vitamin D
- Vitamin D 800 IU (Active Comparator): Group 3 consisted of subjects who were able to receive enteral nutrition, were given antibiotics, and were supplemented with vitamin D3 at a dose of 800 IU once daily for 7 days.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D 400 IU for 7 days
  Other Names: L-VIT D3
  Arms: Vitamin D 400 IU
Drug: Vitamin D — Vitamin D 800 IU for 7 days
  Other Names: L-VIT D3
  Arms: Vitamin D 800 IU

SUMMARY:
The goal of this clinical trial is to learn the effect of vitamin D as an adjunctive therapy for preterm neonates with sepsis measured by the outcomes, which are sepsis score and C-reactive protein after 7 days. The main questions it aims to answer are:

Is there a difference in the results of the sepsis score (Modified Tollner Score and Sepsis Prediction Score) between groups of preterm neonates with sepsis who were given vitamin D as adjuvant therapy at doses of 400 IU/day, 800 IU/day, and those who were only given antibiotics?

Is there a difference in CRP levels between groups of preterm neonates with sepsis who were given vitamin D as adjuvant therapy at doses of 400 IU/day, 800 IU/day, and those who were only given antibiotics?

Participants will be divided into 3 groups:

Group 1 consisted of subjects who were given only antibiotics due to medical conditions requiring fasting.

Group 2 consisted of subjects who were able to receive enteral nutrition, were given antibiotics, and were supplemented with vitamin D3 at a dose of 400 IU once daily for 7 days.

Group 3 consisted of subjects who were able to receive enteral nutrition, were given antibiotics, and were supplemented with vitamin D3 at a dose of 800 IU once daily for 7 days.

DETAILED DESCRIPTION:
The target population in this study is preterm neonates diagnosed with sepsis. This is a multicenter study. The accessible population in this study is patients who are treated in the Neonatal High Care Unit (NHCU) and Neonatal Intensive Care Unit (NICU) at Dr. Hasan Sadikin General Hospital Bandung and Bandung Kiwari Hospital, who meet the inclusion criteria and do not meet the exclusion criteria, and whose parents or guardians are willing to participate in the study by signing the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the case group used in this study are neonates (aged 0-28 days or with a maximum postmenstrual age of 42 weeks) with a gestational age of 28-36 weeks who are treated in the Neonatal High Care Unit (NHCU) and Neonatal Intensive Care Unit (NICU) at Dr. Hasan Sadikin General Hospital, Bandung, and Bandung Kiwari Hospital, Bandung and who meet the following inclusion criteria:

1. Patients diagnosed with neonatal sepsis based on positive blood or cerebrospinal fluid cultures, or who meet the criteria for suspected sepsis with a Rodwell hematologic scoring system result of ≥3.
2. Parents or legal guardians are willing to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Patients with major congenital malformations such as anencephaly, encephalocele, holoprosencephaly, hydrocephalus, meningomyelocele, spina bifida, omphalocele, gastroschisis, or congenital heart disease.
2. If during the 7-day monitoring period, a patient who was initially able to feed develops a medical condition requiring fasting (NPO).
3. If during the 7-day monitoring period, a patient who initially had a medical condition requiring fasting is later able to feed again.

Ages: 0 Days to 84 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2025-08-02 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reni Ghrahani, MD, Ph.D, Study Director — Child Health Department Hasan Sadikin General Hospital Universitas Padjadjaran; Fiva A Kadi, MD, Ph.D, Study Director — Child Health Department Hasan Sadikin General Hospital Universitas Padjadjaran
Locations (2):
- Indonesia (2):
  - Hasan Sadikin General Hospital, Bandung, West Java
  - Rumah Sakit Umum Daerah Bandung Kiwari, Bandung, West Java

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 1 year after the publication of results
Access Criteria: A proposal that describes planned analyses must be submitted and a data sharing agreement must be signed. The proposal must be submitted to the principal investigator's email. The statistical methods for analyses of the proposal must be approved by independent review.

REFERENCES:
- [Background] Fort P, Salas AA, Nicola T, Craig CM, Carlo WA, Ambalavanan N. A Comparison of 3 Vitamin D Dosing Regimens in Extremely Preterm Infants: A Randomized Controlled Trial. J Pediatr. 2016 Jul;174:132-138.e1. doi: 10.1016/j.jpeds.2016.03.028. Epub 2016 Apr 11. PMID 27079965
- [Background] Kamsiah K, Hasibuan BS, Arto KS. The relationship between vitamin D levels and clinical outcomes of neonatal sepsis in Haji Adam Malik Hospital Medan, Indonesia. Open Access Maced J Med Sci. 2021;9(B):698-703.
- [Background] Cetinkaya M, Cekmez F, Buyukkale G, Erener-Ercan T, Demir F, Tunc T, Aydin FN, Aydemir G. Lower vitamin D levels are associated with increased risk of early-onset neonatal sepsis in term infants. J Perinatol. 2015 Jan;35(1):39-45. doi: 10.1038/jp.2014.146. Epub 2014 Aug 7. PMID 25102323
- [Background] Hagag AA, El Frargy MS, Houdeeb HA. Therapeutic Value of Vitamin D as an Adjuvant Therapy in Neonates with Sepsis. Infect Disord Drug Targets. 2020;20(4):440-447. doi: 10.2174/1871526519666190626141859. PMID 31241441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the neonatal intensive care unit (NICU) and neonatal high care unit (NHCU) from 2 medical centers; at a regional hospital and a tertiary care hospital in Bandung, Indonesia, between August 2025 and December 2025
Pre-assignment Details: There were no events or washout periods between participant enrollment and assignment.
Period: Overall Study
Arm/Group | Antibiotics Only | Vitamin D 400 IU | Vitamin D 800 IU
Started | 35 | 20 | 23
Completed | 23 | 19 | 19
Not Completed | 12 | 1 | 4
Not completed — Death | 8 | 0 | 1
Not completed — Achieved enteral nutrition tolerance during monitoring | 4 | 0 | 0
Not completed — Transitioned to nil per os status during monitoring | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotics Only | Vitamin D 400 IU | Vitamin D 800 IU | Total
Number analyzed (Participants) | 23 | 19 | 19 | 61
Age, Customized [Median (Inter-Quartile Range); unit: days]
  Age | 4 [2 to 11] | 10 [5 to 20] | 6 [4 to 13] | 6 [3 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 10 | 28
  Male | 12 | 12 | 9 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gestational Age [Median (Inter-Quartile Range); unit: weeks] | 33 [29 to 34] | 32 [29 to 33] | 32 [32 to 33] | 32 [30 to 34]
Birth Weight [Mean (Standard Deviation); unit: gram] | 1579.5 (568.3) | 1536.7 (386.4) | 1674.3 (397.0) | 1595.7 (462.2)
Respiratory support [Count of Participants; unit: Participants]
  Low flow | 1 | 1 | 1 | 3
  Non-invasive ventilation | 5 | 5 | 6 | 16
  Ventilator | 17 | 13 | 12 | 42
Vitamin D concentration in participants [Median (Inter-Quartile Range); unit: ng/mL] | 9.36 [5.27 to 13.60] | 16.35 [6.64 to 28.30] | 20.50 [8.10 to 24.99] | 11.67 [6.10 to 23.4]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Modified Töllner Sepsis Scoring System After 7 Days
Description: Modified Töllner sepsis scoring system consists of clinical parameters including appearance, microcirculation, hypotonia, bradycardia/tachycardia, apnea of prematurity, respiratory distress, hepatomegaly, gastrointestinal symptoms, leucocyte count, Immature to Total Neutrophil (I/T) ratio, thrombocytopenia, C-reactive protein.
  Minimum value: 0 Maximum value: 26 Higher scores mean a worse outcome for neonatal sepsis
Time Frame: Baseline (day-0) and at day-7
Measure: Median (Inter-Quartile Range); unit: Score
Arm/Group | Antibiotics Only | Vitamin D 400 IU | Vitamin D 800 IU
Number analyzed (Participants) | 23 | 19 | 19
Score
  Day-0 | 7 [6 to 10] | 7 [6 to 9] | 8 [7 to 9]
  Day-7 | 9 [8 to 12] | 2 [0 to 6] | 1 [0 to 6]
  Δ Day 1 and 7 | 1 [0 to 4] | -5 [-7 to -1] | -6 [-8 to -2]
Statistical Analysis 1: Comparison: Antibiotics Only vs Vitamin D 400 IU vs Vitamin D 800 IU; Test type: Superiority; p < 0.001, ANCOVA

2. Primary Outcome: Change From Baseline in the Sepsis Prediction Score After 7 Days
Description: Sepsis Prediction Score consists of clinical parameters including body temperature, decrease feeding volume/residuals, platelet counts, blood glucose changes, C-reactive protein, circulatory changes, increase of oxygen requirement, deterioration of respiratory function.
  Minimum value: 0 Maximum value: 8 Higher scores mean a worse outcome for neonatal sepsis
Time Frame: Baseline (day-0) and at day-7
Measure: Median (Inter-Quartile Range); unit: Score
Arm/Group | Antibiotics Only | Vitamin D 400 IU | Vitamin D 800 IU
Number analyzed (Participants) | 23 | 19 | 19
Score
  Day-0 | 4 [3 to 4] | 3 [2 to 4] | 3 [2 to 4]
  Day-7 | 4 [2 to 5] | 0 [0 to 2] | 0 [0 to 2]
  Δ Day 1 and 7 | 0 [-1 to 1] | -2 [-3 to -1] | -2 [-3 to -1]
Statistical Analysis 1: Comparison: Antibiotics Only vs Vitamin D 400 IU vs Vitamin D 800 IU; Test type: Superiority; p < 0.001, ANCOVA

3. Primary Outcome: Change From Baseline in the C-Reactive Protein Levels After 7 Days
Description: The blood sample was taken from the neonate to test for C-reactive protein (CRP) on day 0 and day 7.
  Minimum value: 0 Higher scores mean a worse outcome for neonatal sepsis
Time Frame: Baseline (day-0) and at day-7
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Antibiotics Only | Vitamin D 400 IU | Vitamin D 800 IU
Number analyzed (Participants) | 23 | 19 | 19
mg/dL
  Day-0 | 0.26 [0.08 to 1.92] | 0.36 [0.13 to 5.93] | 1.19 [0.63 to 11.41]
  Day-7 | 1.71 [0.12 to 9.19] | 0.54 [0.04 to 5.25] | 0.82 [0.19 to 5.82]
  Δ Day 1 and 7 | 0.25 [-0.06 to 4.30] | -0.06 [-4.16 to 1.82] | -0.93 [-7.99 to 0.42]
Statistical Analysis 1: Comparison: Antibiotics Only vs Vitamin D 400 IU vs Vitamin D 800 IU; Test type: Superiority; p = 0.030, ANCOVA

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, up to 7 days
Arm/Group | Antibiotics Only | Vitamin D 400 IU | Vitamin D 800 IU
All-Cause Mortality (participants affected / at risk) | 8/35 | 0/20 | 1/23
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 0/35 | 0/20 | 0/23

LIMITATIONS AND CAVEATS:
Baseline difference: the control group (antibiotic only) consisted solely of neonates kept NPO (nil per os) for medical necessity. In contrast, the intervention groups (vitamin D 400 and 800 IU) were required to be on enteral nutrition. Repeated CRP testing was performed on day 7, although serial monitoring on day 3 is considered ideal. This constraint was due to limitations in blood sampling and laboratory resources at our hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT07245277/Prot_SAP_001.pdf
  • Informed Consent Form (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT07245277/ICF_000.pdf